CLINICAL TRIAL: NCT05920356
Title: A Phase 3, Multicenter, Randomized, Open-label Study Evaluating Efficacy of Sotorasib Platinum Doublet Combination Versus Pembrolizumab Platinum Doublet Combination as a Front-Line Therapy in Subjects With Stage IV or Advanced Stage IIIB/C Nonsquamous Non-Small Cell Lung Cancers, Negative for PD-L1, and Positive for KRAS p.G12C (CodeBreaK 202)
Brief Title: A Study Evaluating Sotorasib Platinum Doublet Combination Versus Pembrolizumab Platinum Doublet Combination as a Front-Line Therapy in Participants With Stage IV or Advanced Stage IIIB/C Nonsquamous Non-Small Cell Lung Cancers (CodeBreaK 202)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190341; 2022-501863-41-00 (EU CTIS Number)
Record Dates: First submitted 2023-05-23; First posted 2023-06-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Oncology; Lung Cancer; PD-L1; KRAS p.G12C; Sotorasib; Pembrolizumab; Carboplatin; Pemetrexed; CodeBreaK 202; NSCLC; PD-L1 Negative; AMG 510; LUMAKRAS ®; LUMYKRAS ®
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Neoplasms | interventions — sotorasib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sotorasib combined with carboplatin and pemetrexed (Experimental): Sotorasib administered in combination with carboplatin and pemetrexed.
  Interventions: Drug: Sotorasib
- Pembrolizumab combined with carboplatin and pemetrexed (Active Comparator): Pembrolizumab administered in combination with carboplatin and pemetrexed.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Sotorasib — Oral administration
  Other Names: AMG 510; LUMYKRAS ®; LUMAKRAS ®
  Arms: Sotorasib combined with carboplatin and pemetrexed
Drug: Pembrolizumab — Intravenous administration
  Arms: Pembrolizumab combined with carboplatin and pemetrexed

SUMMARY:
The primary objectives are to compare progression-free survival (PFS) and overall survival (OS) in participants who receive sotorasib with platinum doublet chemotherapy versus participants who receive pembrolizumab with platinum doublet chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of nonsquamous stage IV or advanced Stage IIIB or IIIC NSCLC with KRAS p. G12C mutation and negative for PD-L1 expression by central testing or local laboratory testing confirmed through central testing
* No history of systemic anticancer therapy in metastatic/non-curable settings
* Eastern Cooperative Oncology Group (ECOG) ≤ 1

Exclusion Criteria:

* Mixed histology NSCLC with either small-cell or large-cell neuroendocrine cell component or predominant squamous cell histology
* Participants with tumors known to harbor molecular alterations for which targeted therapy is locally approved as a front-line therapy
* Symptomatic (treated or untreated) brain metastases
* Gastrointestinal (GI) tract disease causing the inability to take oral medication
* Myocardial infarction within 6 months of randomization, unstable arrhythmias, or unstable angina
* Prior therapy with a KRAS G12C inhibitor

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Approximately 2.5 years
  PFS is defined as the time from randomization until the first documentation of radiologic disease progression or death due to any cause, whichever occurs first. Progression will be based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, per Blinded Independent Central Review (BICR).
Overall Survival (OS) | Approximately 2.5 years
  OS is defined as the time from randomization until death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From Baseline up to end of study (EOS) (approximately 5.5 years)
  Objective response is defined as the best overall response of complete response (CR) or partial response (PR), based on RECIST v1.1, per BICR.
Change in Quality-of-Life Questionnaire Core 30 (QLQ-C30) Dyspnea Domain Score | From Baseline to Week 12
Change in Quality-of-Life Questionnaire Lung Cancer 13 (QLQ-LC13) Symptoms of Dyspnea Subscale | From Baseline to Week 12
Change in QLQ-LC13 Symptoms of Cough Subscale | From Baseline to Week 12
Change in QLQ-LC13 Symptoms of Chest Pain Subscale | From Baseline to Week 12
Change in Physical Function as Measured by QLQ-C30 | From Baseline to Week 12
Change in Global Health Status as Measured by QLQ-C30 | From Baseline to Week 12
Progression-free Survival 2 (PFS2) | From Baseline up to EOS (approximately 5.5 years)
  PFS2 is defined as the time from randomization to progression per investigator after initiation of new anticancer therapy or death from any cause, whichever occurs first.
Change in QLQ-LC13 Subscale Scores | From Baseline up to EOS (approximately 5.5 years)
Change in QLQ-C30 Subscale Scores | From Baseline up to EOS (approximately 5.5 years)
Time to Deterioration in QLC-LC13 Subscale Scores | From Baseline to Week 12
Time to Deterioration in QLC-C30 Subscale Scores | From Baseline to Week 12
Change in Summary Scores and Visual Analogue Scale (VAS) Scores | From Baseline up to EOS (approximately 5.5 years)
  Measured by EuroQol-5 Dimension (EQ-5D-5L).
Duration of Response | From Baseline up to EOS (approximately 5.5 years)
  Duration of response is defined as the time from the first documentation of objective response until the first documentation of disease progression per BICR or death due to any cause, whichever occurs first.
Time to Response | From Baseline up to EOS (approximately 5.5 years)
  Defined as the time from randomization to first evidence of PR or CR per BICR.
Disease Control | From Baseline up to EOS (approximately 5.5 years)
  Defined as CR plus PR plus stable disease based on RECIST v1.1 per BICR.
PFS | From Baseline up to EOS (approximately 5.5 years)
  Based on investigator tumor assessments per RECIST v1.1.
Objective Response | From Baseline up to EOS (approximately 5.5 years)
  Based on investigator tumor assessments per RECIST v1.1.
Number of Participants With Treatment-Emergent Adverse Events | From Baseline up to EOS (approximately 5.5 years)
Number of Participants With Clinically Significant Changes in Vital Signs | From Baseline up to EOS (approximately 5.5 years)
Number of Participants With Clinically Significant Changes in Clinical Laboratory Tests | From Baseline up to EOS (approximately 5.5 years)
Maximum Plasma Concentration (Cmax) of Sotorasib | Pre-dose Day 1 up to Day 64
Minimum Plasma Concentration (Cmin) of Sotorasib | Pre-dose Day 1 up to Day 64
Area Under The Curve (AUC) of Sotorasib | Pre-dose Day 1 up to Day 64

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (377):
- United States (18):
  - Sansum Clinic, Santa Barbara, California
  - Medical Oncology Hematology Consultants Helen F Graham Cancer Center, Newark, Delaware
  - University of Illinois Chicago, Chicago, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Norton Cancer Institute - Brownsboro, Louisville, Kentucky
  - Reliant Medical Group Inc, Worcester, Massachusetts
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - FirstHealth Cancer Center, Pinehurst, North Carolina
  - Alliance Cancer Specialists - Media, Media, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Tennessee Medical Center Knoxville, Knoxville, Tennessee
  - Regional One Health, Memphis, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - United States Oncology Regulatory Affairs Corporate Office, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - US Oncology Research Investigational Products Center, Irving, Texas
- Argentina (10):
  - Hospital Britanico de Buenos Aires, CABA, Buenos Aires
  - Instituto Alexander Fleming, Capital Federal, Buenos Aires
  - Instituto Argentino de Diagnostico y Tratamiento IADT, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Fundacion Ars Medica, San Salvador de Jujuy, Jujuy Province
  - Clinica Viedma, Viedma, Río Negro Province
  - Sanatorio Parque SA, Rosario, Santa Fe Province
  - Centro Oncologico Korben, Buenos Aires
  - Fundacion Centro Oncológico Riojano Integral para la Investigación y Prevención del Cáncer, La Rioja
  - Centro de Diagnostico Investigacion y Tratamiento, Salta
- Australia (11):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Nepean Cancer Centre, Kingswood, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - GenesisCare -North Shore Oncology, St Leonards, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Toowoomba Hospital, Toowoomba, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Cancer Research South Australia, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Austria (5):
  - Medizinische Universitaet Graz, Graz
  - Klinikum Klagenfurt am Woerthersee, Klagenfurt
  - Universitaetsklinikum Krems, Krems
  - Landeskrankenhaus Salzburg, Salzburg
  - Klinikum Wels - Grieskirchen GmbH, Wels
- Belgium (5):
  - Chirec - Delta Ziekenhuis, Auderghem
  - Algemeen Ziekenhuis Maria Middelares, Ghent
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Regional de la Citadelle, Liège
  - Algemeen Ziekenhuis Sint Maarten-Emmaus vzw, Mechelen
- Brazil (21):
  - Hospital Evangelico de Cachoeiro de Itapemirim, Cachoeiro de Itapemirim, Espírito Santo
  - Núcleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Hospital Sirio Libanes Brasilia, Brasília, Federal District
  - Oncoclinicas Onco Vida Distrito Federal, Brasília, Federal District
  - Nucleo de Ensino Pesquisa e Inovacao Mario Penna, Belo Horizonte, Minas Gerais
  - Centro de Tratamento Oncologico - Cto, Belém, Pará
  - Instituto Medicina Integral Imip, Recife, Pernambuco
  - Liga Norte-Riograndense Contra O Cancer, Natal, Rio Grande do Norte
  - Associação Beneficente de Canoas, Canoas, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Centro de pesquisa em oncologia Hospital Ana Nery, Santa Cruz do Sul, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Fundacao pio xII Barretos, Barretos, São Paulo
  - Santa Casa de Misericordia de Santos - Iscms, Santos, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Beneficencia Portuguesa de Sao Paulo - Bp, São Paulo, São Paulo
  - Fundacao Antonio Prudente, São Paulo, São Paulo
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
  - Instituto de Ensino e Pesquisa Sao Lucas Iep Sao Lucas, São Paulo
  - Instituto Cancer Sao Paulo Icesp, São Paulo
- Bulgaria (5):
  - Multiprofile Hospital for Active Treatment - Uni Hospital OOD, Panagyurishte
  - University Multiprofile Hospital for Active Treatment Sveta Marina - Pleven OOD, Pleven
  - Multiprofile Hospital for Active Treatment for Womens Health - Nadezhda OOD, Sofia
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment Tokuda EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
- Canada (7):
  - Queen Elizabeth II, Health Sciences Centre, Halifax, Nova Scotia
  - Sunnybrook Research Institute Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill University Health Centre Glen Site, Montreal, Quebec
  - CIUSSS - du Nord-de-lIle-de-Montreal / Hopital Sacre-Coeur de Montreal, Montreal, Quebec
  - Institut Universitaire de cardiologie et de pneumologie de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Chile (6):
  - James Lind Centro de Investigacion del Cancer, Temuco, Cautín
  - Clinica CIDO, Temuco, Cautín
  - Orlandi Oncologia, Santiago
  - Fundacion Arturo Lopez Perez, Santiago
  - Biocinetic servicios medicos limitada, Santiago
  - Centro de Investigacion del Maule, Talca
- China (50):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Anhui Chest Hospital, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Gansu Province Cancer Hospital, Lanzhou, Gansu
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Affiliated Cancer Hospital and institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Liuzhou Peoples Hospital, Liuchow, Guangxi
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Hainan Cancer Hospital, Haikou, Hainan
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - AnYang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science And Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College Of Hust, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Linyi Peoples Hospital, Linyi, Shandong
  - Weifang Peoples Hospital, Weifang, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi An JiaoTong University, Xi’an, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - the First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Nantong Tumor Hospital, Nantong, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital, Capital Medical University, Beijing
- Colombia (8):
  - Fundacion Colombiana de Cancerologia Clinica Vida, Medellín, Antioquia
  - Sociedad de Oncologia y Hematologia del Cesar, Valledupar, Cesar Department
  - Instituto Nacional de Cancerologia, Bogota, Cundinamarca
  - Centro de Tratamiento e Investigación sobre Cancer Luis Carlos Sarmiento Angulo Ctic, Bogotá, Cundinamarca
  - Instituto Medico de Alta Tecnologia sas - Imat sas, Montería, Departamento de Córdoba
  - Oncologos del Occidente SAS, Pereira, Risaralda Department
  - Fundacion cardiovascular de Colombia, Bucaramanga, Santander Department
  - Centro Cancerologico del Caribe LTDA CECAC, Barranquilla
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Plzen, Pilsen
- Denmark (5):
  - Aarhus Universitetshospital, Aarhus N
  - Rigshospitalet, Copenhagen
  - Regionshospitalet Godstrup, Herning
  - Sonderborg Sygehus, Sønderborg
  - Vejle Sygehus, Vejle
- France (29):
  - Centre Hospitalier Regional Universitaire de Besancon - Hopital Jean Minjoz, Besançon
  - Centre Hospitalier Universitaire Ambroise Pare, Boulogne-Billancourt
  - Centre Hospitalier Universitaire de Caen - Hopital Cote de Nacre, Caen
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Centre Hospitalier Departemental Les Oudairies, La Roche-sur-Yon
  - Centre Hospitalier - Le Mans, Le Mans
  - Centre Hospitalier Régional Universitaire de Lille - Institut Coeur Poumon, Lille
  - Centre Hospitalier Universitaire Nord, Marseille
  - Centre de Cancerologie du Grand Montpellier-Clinique Clementville, Montpellier
  - Hopital prive du Confluent, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hopital Universitaire Caremeau, Nîmes
  - Institut Curie, Paris
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - Hopital Cochin, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Universitaire de Poitiers - Hopital la Miletrie, Poitiers
  - Centre Hospitalier de Cornouaille, Quimper
  - Centre Hospitalier Universitaire de Reims - Hopital Christian Cabrol, Reims
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Rouen - Hopital Charles Nicolle, Rouen
  - Centre Hospitalier Universitaire de Saint Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - Centre Hospitalier Universitaire de Strasbourg - Nouvel Hopital Civil, Strasbourg
  - Hopital d instruction des armees sainte anne, Toulon
  - Centre Hospitalier Universitaire de Toulouse - Hopital Larrey, Toulouse
  - Centre Hospitalier Regional Universitaire de Tours - Hopital Bretonneau, Tours
  - Hopital Nord Ouest Villefranche sur Saone, Villefranche-sur-Saône
  - Gustave Roussy, Villejuif
- Germany (5):
  - Klinikum Chemnitz GmbH, Chemnitz
  - Asklepios Fachkliniken Muenchen Gauting, Gauting
  - Universitaetsmedizin Goettingen, Göttingen
  - Klinikverbund Allgaeu, Kempten
  - Klinikum der LMU Muenchen, München
- Greece (11):
  - 251 General Airforce Hospital, Athens
  - Henry Dunant Hospital Center, Athens
  - Alexandra Hospital, Athens
  - Attikon University Hospital, Athens
  - Iaso Hospital, Athens
  - Metropolitan Hospital, Athens
  - Iaso General Clinic, Marousi
  - Metaxa Anticancer Hospital, Piraeus
  - Theagenion Cancer Hospital, Thessaloniki
  - Agios Loukas Clinic, Thessaloniki
  - European Interbalkan Medical Center, Thessaloniki
- Hong Kong (3):
  - Queen Mary Hospital, The University of Hong Kong, Hong Kong
  - Princess Margaret Hospital, Kowloon
  - Queen Elizabeth Hospital, Hong Kong, Kowloon
- Hungary (9):
  - Orszagos Koranyi Pulmonologiai Intezet, Budapest
  - Budapesti Uzsoki Utcai Korhaz, Budapest
  - Farkasgyepui Tudogyogyintezet, Farkasgyepű
  - Matrai Gyogyintezet, Gyöngyös
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktatokorhaz, Győr
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - Jasz-Nagykun-Szolnok Varmegyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
  - Komarom-Esztergom Varmegyei Szent Borbala Korhaz, Tatabánya
  - Reformatus Pulmonologiai Centrum, Törökbálint
- Italy (14):
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - Azienda Socio Sanitaria Territoriale Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero Universitaria Policlinico G Rodolico - San Marco Presidio Ospedaliero G Rodolico, Catania
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori, Meldola (FC)
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza (MB)
  - Azienda Ospedaliera di Rilievo Nazionale Specialistica dei Colli Monaldi, Napoli
  - Azienda Ospedaliero Universitaria Luigi Vanvitelli, Napoli
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Azienda Ospedaliera di Perugia Ospedale Santa Maria della Misericordia, Perugia
  - Azienda Sanitaria Territoriale Pesaro Urbino - Presidio San Salvatore Muraglia, Pesaro
  - IRCCS Istituti Fisioterapici Ospitalieri, Rome
  - Azienda Sanitaria Universitaria Friuli Centrale Presidio Ospedaliero Santa Maria della Misericordia, Udine
- Japan (32):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hirosaki University Hospital, Hirosaki-shi, Aomori
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Ehime University Hospital, Toon-shi, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Japan, Kitakyushu-shi, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Chugoku Central Hospital of Japan Mutual Aid Association of Public School Teachers, Fukuyama-shi, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kobe Minimally invasive Cancer Center, Kobe, Hyōgo
  - Takarazuka City Hospital, Takarazuka-shi, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - St Marianna University Hospital, Kawasaki-shi, Kanagawa
  - Kanagawa Prefectural Hospital Organization Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kyoto University Hospital, Kyoto, Kyoto
  - Miyagi Cancer Center, Natori-shi, Miyagi
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Sakai-shi, Osaka
  - National Hospital Organization Kinki-chuo Chest Medical Center, Sakai-shi, Osaka
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - Tottori University Hospital, Yonago-shi, Tottori
  - Wakayama Medical University Hospital, Wakayama, Wakayama
  - National Hospital Organization Yamaguchi-Ube Medical Center, Ube-shi, Yamaguchi
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East Clinical University Hospital, Riga
- Malaysia (3):
  - Pantai Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
- Mexico (6):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Health Pharma Professional Research SA de CV, Mexico City, Mexico City
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Oncare, Monterrey, Nuevo León
  - Actualidad Basada en la Investigación del Cáncer, Guadalajara
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
- Netherlands (6):
  - Meander Medisch Centrum, Amersfoort
  - Universitair Medisch Centrum Groningen, Groningen
  - Sint Jansdal Ziekenhuis, Harderwijk
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
  - Isala Klinieken, Zwolle
- Peru (5):
  - Centro de Investigacion Vallesur, Arequipa
  - Hospital Nacional Adolfo Guevara Velasco, Cusco
  - Oncosalud, Lima
  - Unidad de Investigación Clínica Internacional Sede San Borja, Lima
  - Hospital de Apoyo Departamental Maria Auxiliadora, Lima
- Poland (10):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Centrum Pulmonologii i Torakochirurgii w Bystrej, Bystra
  - Szpitale Pomorskie spolka z ograniczona odpowiedzialnoscia, Gdynia
  - Szpital Specjalistyczny imienia Ludwika Rydygiera w Krakowie Sp zoo, Krakow
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Uniwerystecki Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Med Polonia Sp zoo, Poznan
  - Wojewodzki Szpital im Sw Ojca Pio w Przemyslu, Przemyśl
  - Narodowy Instytut Onkologii im Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw
  - Specjalistyczny Szpital im Dra Alfreda Sokolowskiego, Wałbrzych
- Portugal (6):
  - Hospital Cuf Tejo, Lisbon
  - Fundacao Champalimaud, Lisbon
  - Hospital da Luz, SA, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE - Hospital Pulido Valente, Lisbon
  - Unidade Local de Saude de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - Hospital Cuf porto, Porto
- Romania (8):
  - Institutul Oncologic, Prof Dr Alexandru Trestioreanu, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - SC Medisprof SRL, Cluj-Napoca
  - Centrul de Oncologie Sf Nectarie SRL, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Municipal Ploiesti, Ploieşti
  - SC Oncomed SRL, Timișoara
- Singapore (2):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (8):
  - Pusan National University Hospital, Busan
  - National Cancer Center, Goyang-si Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan-si, Gyeongsangnam-do
- Spain (17):
  - Hospital Regional Universitario de Malaga, Málaga, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Institut Catala d Oncologia Hospitalet Hospital Duran i Reynals, L'Hospitalet de Llobregat, Catalonia
  - Complexo Hospitalario Universitario A Coruna Hospital Teresa Herrera, A Coruña, Galicia
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
- Sweden (3):
  - Gavle Sjukhus, Gävle
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Norrlands Universitetssjukhus, Umeå
- Switzerland (4):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital Basel, Basel
  - Universitaetsspital Zuerich, Zurich
- Taiwan (7):
  - China Medical University Hospital, Taichung
  - Veterans General Hospital - Taichung, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital, Liouying, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Thailand (7):
  - Vajira Hospital, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Banphaeo General Hospital, Samut Sakhon
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (18):
  - Medical Park Seyhan Hastanesi, Adana
  - Baskent Universitesi Adana Doktor Turgut Noyan Uygulama ve Arastirma Merkezi, Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Gazi Universitesi Saglik Arastirma ve Uygulama Merkezi Gazi Hastanesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Aydin Adnan Menderes Universitesi Tip Fakultesi, Aydin
  - Pamukkale Universitesi Tip Fakultesi Hastanesi, Denizli
  - Prof Dr Cemil Tascioglu Sehir Hastanesi, Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Memorial Bahcelievler Hastanesi, Istanbul
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - Goztepe Prof Dr Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Kartal Dr Lutfi Kirdar Sehir Hastanesi, Istanbul
  - Marmara Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Dr Suat Seren Gogus Hastaliklari ve Cerrahisi Egitim ve Arastirma Hastanesi, Izmir
  - Izmir Ekonomi Universitesi Medical Point Hastanesi, Izmir
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
- United Kingdom (8):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Raigmore Hospital, Inverness
  - Royal Marsden Hospital, London
  - Mount Vernon Cancer Centre, Northwood
  - Nottingham City Hospital, Nottingham
  - Royal Marsden Hospital, Sutton
  - Torbay Hospital, Torquay
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com